CLINICAL TRIAL: NCT01567254
Title: Subject: A Blinded Randomized Trial: the Effect of Guided Imagery in Children With Type 1 Diabetes Mellitus on Glucose Levels and on Glycemic Control
Brief Title: The Effect of Guided Imagery in Children With Type 1 Diabetes Mellitus on Glucose Levels and on Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Dr. Marianna Rachmiel, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 54/11
Record Dates: First submitted 2012-02-01; First posted 2012-03-30 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
Keywords: guided imaginary
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- guided imaginary (Experimental): 7 children receiving auditory guided imagery disk
  Interventions: Behavioral: guided imaginary
- music (Active Comparator): 6 children receiving music disk
  Interventions: Behavioral: music ONLY

INTERVENTIONS:
Behavioral: guided imaginary — Auditory guided imagery disk - will be prepared by Ronit Brooks, a clinical psychologist, who is engaged in guided imagery and by Livia Yanai, an art therapist.
  Other Names: N\A
  Arms: guided imaginary
Behavioral: music ONLY — music. It will be equal in length to the auditory guided imagery disk
  Other Names: N\A
  Arms: music

SUMMARY:
Background: Pediatric patients with type 1 diabetes mellitus are known to be a challenging group for achieving recommended glycemic control. Coping with the demands of self-managing IDDM in children and adolescents can be a formidable task, requiring a healthy and balanced diet, monitoring and regular insulin injections. Most patients are non-compliant to the treatment. A number of controlled studies have examined the efficiency of psychosocial interventions for improving compliance and glycemic control among diabetic youth. None has examined the effectiveness of guided imagery in treatment of type 1 diabetes mellitus.

Primary Objective: To asses simultaneously the effect of listening to auditory guided imagery and blood glucose variability, compared to variability in blood glucose while listening to songs.

Secondary Objective To assess the effect of routine auditory guided imagery to glycemic control and quality of life in children with type 1 diabetes mellitus, compared to listening listening to songs.

Methods:

Subjects: 14 youth ages 7-16 years with type 1 diabetes mellitus , for at least 6 months, and not during the honey moon period will be recruited, and will be blindly randomized to receive intervention (auditory guided imagery group) or control (regular auditory music).

Protocol:

Design: A randomized Controlled Blinded Study Intervention: 14 randomly numbered CD's will be prepared at study initiation, half containing auditory guided imagery and half containing music.

Study protocol: After an initial check up, including HbA1C levels, and explanation of study procedures the participants will be given either the intervention or the control CD, to be used twice a day for five days. During this period continuous glucose monitoring will be performed. On days one and five the procedure will take place while the participants are connected to biofeedback. QOL questionnaires will be completed at the beginning of day one, or before.

In the second part of the study the children will use the intervention / control CD at home twice a week for 12 weeks. At the end of the study period they will again be evaluated, including HbA1C, and all subjects will again complete QOL questionnaires

DETAILED DESCRIPTION:
14 participants will be assigned research numbers in a consecutive recruitment order.(01-14).

14 auditory disks will be prepared ahead of study initiation, 7 with the guided imagery program and 7 with regular songs.

All will look similar from the outside. The disks will be numbered 01-14. Disks numbering will be performed by an investigator who is not part of treatment team, without knowing which disk contains which content. So that the team and participants are blinded to the disk content at initiation.

Children and parents will be aware of the type of auditory disk after initial auscultation at visit number 1.

The team will continue to be blinded to type of disk until end of study. 3. All participants will be aware at study initiation that they may receive the auditory guided imagery disk or a regular songs / story auditory disk.

4. Visit no. 1:

1. Will be arranged on date of their regular clinic visit
2. Guidance to disk usage
3. Biofeedback for autonomic parameters assessment
4. Participants will be connected to the continuous glucose monitoring system (A system which the patient is blinded to glucose readings).
5. Participants and parents will fill QOL questionnaire [The Diabetes Treatment Satisfaction Questionnaire (DTSQ) by Bradley C. et Al (16)], if not filled before.
6. Participants will listen to disk for the first time in clinic, alone in a room with the parent
7. At this stage participants will be aware of the group they are in (treatment vs. control), but team is still unaware.
8. Participants will be able to come with brothers and parents and recreational activity will be available at site for all for entertainment 5. Visit no. 2-5: 6. Participants will listen to disk twice a day for the next four days alone in a room in our clinic. They will be able to come with brothers and parents, and recreational activity will be available at site for all for entertainment.

   7. 5th day visit:

a. Participants will listen to disk for the last times in clinic, alone in a room.

b. Participants will be disconnected from CGMS c. Biofeedback for autonomic parameters assessment 8. Participants will listen to disk at least twice a week, for additional 11 weeks, at their choice of time and day, and will record the specific time of listening on study chart 9. Visit no. 6:

1. Will be arranged on date of their regular clinic visit (12-14 weeks after visit no. 1)
2. Biofeedback for autonomic parameters assessment
3. Participants and parents will fill QOL questionnaires (The Diabetes Treatment Satisfaction Questionnaire (DTSQ) by Bradley C. et Al (16)
4. End of study 10. Data will be collected from charts from dates of visit no. 1 and visit no. 3 regarding: weight, height, BMI, 14 days average blood glucose levels, HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for longer than 6 months
* Insulin requirements of more than 0.4 units/kg/day for at least 3 months
* Age 7-16 years
* Agreement of parents or guardian to participate in the study
* Agreement and wiliness of child to participate in the study

Exclusion Criteria:

* Children with cognitive impairment which prevents them from using guided imagery
* Unable to understand Hebrew
* Hearing defect
* Attention deficit disorder

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Blood glucose values before and after listening to the recording. | 1 week
  Blood glucose variability of teenagers before and after listening to auditory guided imagery, compared to the blood glucose variability of teenagers before and after listening to music. The blood glucose values will be measured by continuous glucose monitoring system (CGMS).

SECONDARY OUTCOMES:
The delta of HA1C between before and after three months of periodic listening to auditory guided imagery, compared to listening to music. | 3 months
  Average of deltas of HA1C between before and after three months of peridic listening to auditory guided imagery, compared to listening to music.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Rachmiel, MD, Principal Investigator — Hassaf Haroffeh Medical Center
Locations (1):
- Assaf Haroffeh Medical center, Ẕerifin, Israel